CLINICAL TRIAL: NCT03742856
Title: A Multi-omics Study on the Invasiveness of Epithelial Ovarian Cancer
Brief Title: A Multi-omics Study of Epithelial Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-OMICS
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Epithelial Ovarian Cancer; Tumor Invasiveness; Whole Exome Sequencing; Transcriptomics; Metabolomics; Tumorigenesis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An 8 ml peripheral venous blood, and 50 μL cancer tissue and tissue adjacent to cancer will be collected from eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: A multi-omics analysis — A multi-omics analysis including whole exome sequencing, transcriptomics and metabolomics.

SUMMARY:
This study aims to analyze the multi-omics results between epithelial ovarian cancer (EOC) patient with different FIGO stages and pathological subtypes. The multi-omics profiles include whole exome sequencing, analysis of transcriptomics and metabolomics. A comprehensive multi-omics will reveal the invasiveness and tumorigenesis of EOC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary epithelial ovarian cancer
* Signed an approved informed consents
* Feasible for biopsy

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients confirmed primary epithelial ovarian cancer will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-11-23 (Estimated); Study Completion 2020-11-23 (Estimated)

PRIMARY OUTCOMES:
Frequencies of somatic driving mutations | Two years
  The differences of frequencies of somatic driving mutations will be compared between patients of different FIGO stages and different pathological subtypes.

SECONDARY OUTCOMES:
Frequencies of alteration of RNA expression | Two years
  The alteration of RNA expression, including mRNA, miRNA, and lncRNA, will be compared between patients of different FIGO stages and different pathological subtypes.
Frequencies of alteration of protein expression and signal pathway | Two years
  The alteration of patterns of protein expression and signal pathway will be compared between patients of different FIGO stages and different pathological subtypes.
Progression-free survival | Five years
  Progression-free survival between patients with differential expressed multi-omics will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China